CLINICAL TRIAL: NCT03344978
Title: Cardboard Cot in Neonatal Thermoregulation: A Randomized Cross Over Trial in Prevention of Moderate or Severe Hypothermia in Preterm Infants Requiring at Least 1 Week of Incubator
Brief Title: Cardboard Cot in Neonatal Thermoregulation: A Randomized Cross Over Trial
Acronym: CCot
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit participants
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Colm Travers, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: UAB Neo 018
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Infant, Premature; Hypothermia, Newborn
Keywords: Neonate; Premature; Hypothermia; Cardboard; Cot
MeSH Terms: conditions — Premature Birth; Hypothermia

STUDY DESIGN:
Intervention Model Description: Randomized crossover. Participant will be randomly assigned initially to care in one of two devices for 24 hours, then crossed over to other device for 24 hours. This will be repeated once more for a total of 96 hours study time. Patterns may be A-B-A-B or B-A-B-A.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardboard Cot Care (Active Comparator): Stable infant will be nursed in a cardboard cot, lined with reflective film for 24 hour period of time. Infant's axillary temperature will be taken at 1 hour after randomization, at 6 hours after randomization, and 24 hours after randomization. After 24 hours, infant will be swapped to the other arm (Incubator Care), and back for a total of 2 24-hour periods in each arm.
  Interventions: Other: Cardboard Cot Care
- Incubator Care (Placebo Comparator): Stable infant will be nursed in an incubator for 24 hour period of time. Infant's axillary temperature will be taken at 1 hour after randomization, at 6 hours after randomization, and 24 hours after randomization. After 24 hours, infant will be swapped to the other arm (Cardboard Cot Care), and back for a total of 2 24-hour periods in each arm.
  Interventions: Other: Incubator Care

INTERVENTIONS:
Other: Cardboard Cot Care — Infant maintained in reflective film-lined cot for a period of 24 hours. Axillary temperatures will be taken at 1 hour, 6 hours, and 24 hours after randomization. If temperatures found < 36° C. at any time, an additional blanket and hat will be added to infant to improve temperature. Infant may be moved to incubator or radiant warmer. All other care will be standard of care at University Teaching Hospital, including warm delivery rooms, immediate drying, postponed bathing and weighing, early and exclusive breastfeeding, and Kangaroo Mother Care as continuously as possible.
  Other Names: CCot
  Arms: Cardboard Cot Care
Other: Incubator Care — Infant maintained in standard incubator for a period of 24 hours. Axillary temperatures will be taken at 1 hour, 6 hours, and 24 hours after randomization. If temperatures found < 36° C. at any time, an additional blanket and hat will be added to infant to improve temperature. All other care will be standard of care at University Teaching Hospital, including warm delivery rooms, immediate drying, postponed bathing and weighing, early and exclusive breastfeeding, and Kangaroo Mother Care as continuously as possible.
  Arms: Incubator Care

SUMMARY:
This study will determine whether the efficacy of Mylar-lined cardboard cots is equivalent to traditional incubators in their ability to prevent hypothermia (axillary temperature < 36° C) in preterm neonates <36 6/7 weeks gestational age in a randomized cross-over designed trial. Infants will be randomized to receive care in the cardboard cot or incubator and then cross over to the other device for 24 hour periods, rotating for a total of 96 hours total trial time.

DETAILED DESCRIPTION:
The aim of the trial is to determine whether a corrugated cardboard cot will assist in maintaining infant axillary temperatures comparing it to the temperatures of the same infant being nursed in low heat incubators. The study will be done in the context of standard medical care, including the WHO thermoregulation protocol (warm delivery rooms, immediate drying after birth, early and exclusive breastfeeding, postponement of bathing and weighing, and appropriate bundling).

The cardboard cot is approximately 24 inches long to accommodate the length of the infant and about 12 inches wide to accommodate term infants, even beyond the first months after birth. The cots are fully lined with a reflective metallized film sheet of Mylar. The cot will be covered with a cardboard piece also lined in reflective film up to about the infant's shoulders so that the infant's face is visible. Attached to the lid is a 5 inch cardboard flap lined with reflective film which folds down into the body of the cot to reduce heat loss.

Infants ≤ 36 6/7 weeks gestation will be randomized to receive care in a cardboard cot or an incubator. Infants will begin care in one device and after 24 hours will cross over to the other device for another 24 hours. The process will be repeated once more for a total of 96 hours of study duration. The infants will be normothermic and stable when they are enrolled in the trial. Axillary temperatures will be measured at 1 hr, 6 hours and 24 hours after being placed in the cost or incubator. Infants with observed hypothermia (<36° C) will have measures taken to increase temperature (i.e. adding blankets, hat).

ELIGIBILITY:
Inclusion Criteria:

* Estimated gestational age < 36 6/7 weeks
* Hospitalized in the NICU at University Teaching Hospital in Zambia
* Requiring incubator/radiant warmer for at least 1 week

Exclusion Criteria:

* Abdominal wall defect or myelomeningocele
* Major congenital anomalies
* Blistering skin disorder
* Suspected Sepsis
* Requiring ongoing respiratory support

Ages: 1 Minute to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Moderate (32.-35.9° C) or Severe (<32.0° C) hypothermia per Axillary Temperature | 1 hour after placement in warming device
  Temperature taken via axilla for 1 minute duration
Moderate (32.0-35.9° C) or Severe (<32.0° C) hypothermia per Axillary Temperature | 6 hours after placement in warming device
  Temperature taken via axilla for 1 minute duration
Moderate (32.-35.9° C) or Severe (<32.0°C) hypothermia per Axillary Temperature | 24 hours after placement in warming device
  Temperature taken via axilla for 1 minute duration

SECONDARY OUTCOMES:
Normothermia (Axillary temperature 36.0 - 38.0° C) | 1-96 hours after beginning of study
  Temperature taken via axilla for 1 minute duration
Hypothermia (Axillary temperature < 36.0° C) | 1-96 hours after beginning of study
  Temperature taken via axilla for 1 minute duration
Mean Axillary Temperature in each device | 4 months
  Average of all axillary temperatures taken per device
Rate of Moderate hypothermia (32.0-35.9° C) after placement in warming device | 1 hour after placement in warming device
  Temperature taken via axilla for 1 minute duration
Rate of Moderate hypothermia (32.0-35.9°C) after placement in warming device | 6 hours after placement in warming device
  Temperature taken via axilla for 1 minute duration
Rate of Moderate hypothermia (32.0-35.9° C) after placement in warming device | 24 hours after placement in warming device
  Temperature taken via axilla for 1 minute duration
Rate of Severe hypothermia (<32.0° C) after placement in warming device | 1 hour after placemnt in warming device
  Temperature taken via axilla for 1 minute duration
Rate of Severe hypothermia (<32.0° C) after placement in warming device | 6 hours after placement in warming device
  Temperature taken via axilla for 1 minute duration
Rate of Severe hypothermia (<32.0° C) after placement in warming device | 24 hours after placement in warming device
  Temperature taken via axilla for 1 minute duration
Rate of Hyperthermia (>38.0°C) after placement in warming device | 4 months
  Temperature taken via axilla for 1 minute duration

CONTACTS AND LOCATIONS:
Overall Officials: Colm P Travers, MB BCh BAO, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No